CLINICAL TRIAL: NCT03815747
Title: MRI Evaluation of Change in Gluteal Muscles Following the Treatment With HIFEM Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-799-MRI
Record Dates: First submitted 2019-01-22; First posted 2019-01-24 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Muscle Tone Increased
MeSH Terms: conditions — Muscle Hypertonia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment Group (Experimental): Treatment with the investigational device - High- Intensity Focused Electromagnetic (HIFEM) Field Device
  Interventions: Device: High-Intensity Focused Electromagnetic (HIFEM) Field Device

INTERVENTIONS:
Device: High-Intensity Focused Electromagnetic (HIFEM) Field Device — The High-Intensity Focused Electromagnetic (HIFEM) Field device will be applied.

SUMMARY:
This study will use magnetic resonance imaging (MRI) to evaluate changes in gluteal muscle following the treatment with HIFEM stimulation for aesthetic improvement of buttocks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years
* Voluntarily signed informed consent form
* BMI ≤ 30 kg/m2
* Women of child-bearing potential are required to use birth control measures during the whole duration of the study
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure to promote body contouring during study participation
* Subjects willing and able to maintain his/her regular (pre-procedure) diet and exercise regimen without effecting significant change in either direction during study participation

Exclusion Criteria:

* Cardiac pacemakers
* Implanted defibrillators, implanted neurostimulators
* Electronic implants
* Pulmonary insufficiency
* Metal implants
* Drug pumps
* Malignant tumor
* Fever
* Pregnancy
* Breastfeeding
* Following recent surgical procedures when muscle contraction may disrupt the healing process
* Application over areas of the skin which lack normal sensation
* Scars, open lesions and wounds at the treatment area
* Unrepaired abdominal hernia

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the device for toning of buttocks according to MRI images | 7 months
  Evaluation of change in MRI images before and after the therapy procedure.

SECONDARY OUTCOMES:
Subject's satisfaction with study treatment | 7 months
  Subject's satisfaction with the therapy results evaluated through the Subject Satisfaction Questionnaire. The 7-point Likert scale Subject Satisfaction Questionnaire will be used for an analysis of the subject's opinion of the therapy results.
Side effects and adverse events (AE) associated with the study device | 7 months
  The occurrence of side effects and adverse events will be followed throughout the whole study

CONTACTS AND LOCATIONS:
Locations (1):
- Art of Skin MD, Solana Beach, California, United States